CLINICAL TRIAL: NCT03136458
Title: Efficacy of Remote Ischemic Preconditioning as Non Pharmacologic Strategy to Prevent Contrast Induced Nephropathy (PAIR Trial)
Brief Title: Efficacy of Remote Ischemic Preconditioning as Non Pharmacologic Strategy to Prevent Contrast Induced Nephropathy (PAIR)
Acronym: PAIR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No resources
Sponsor: Camilo Andrés Páez Angarita (Other)
Responsible Party: Sponsor-Investigator, Camilo Andrés Páez Angarita, Internal Medicine Resident, Fundacion Clinica Valle del Lili
Organization: Fundacion Clinica Valle del Lili (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ValledelLili
Record Dates: First submitted 2017-04-24; First posted 2017-05-02 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Contrast-induced Nephropathy
Keywords: contrast media; nephropathy; ischemic preconditioning
MeSH Terms: conditions — Kidney Diseases | interventions — Ischemic Preconditioning

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real ischemic preconditioning (Experimental): Insufflation of an arterial pressure cuff located in one upper extremity, during 4 cycles, each with a duration of 5 minutes insufflation and 5 minutes of disinflation. The cuff will be insufflated to reach 50 mmHg above the systolic arterial pressure of the patient.
  Interventions: Procedure: Ischemic preconditioning; Drug: Endovenous normal saline
- Dummy ischemic preconditioning (Active Comparator): Insufflation of an arterial pressure cuff located in one upper extremity, during 4 cycles, each with a duration of 5 minutes insufflation and 5 minutes of disinflation. The cuff will be insufflated to reach 10 mmHg above the diastolic arterial pressure of the patient.
  Interventions: Drug: Endovenous normal saline

INTERVENTIONS:
Procedure: Ischemic preconditioning — Repeated remote ischemic preconditioning by arterial cuff insufflation.
  Other Names: remote ischemic preconditioning
  Arms: Real ischemic preconditioning
Drug: Endovenous normal saline — endovenous normal saline 1 mL per Kg per hour before and after contrast media injection.
  Other Names: normal saline 0,9%

SUMMARY:
This study evaluates remote ischemic preconditioning as an strategy to avoid contrast induced nephropathy. All of the patients will receive endovenous normal saline to prevent nephropathy, half of the patients will receive remote ischemic preconditioning while the other half will not.

DETAILED DESCRIPTION:
This study evaluates remote ischemic preconditioning as an strategy to avoid contrast induced nephropathy, this preconditioning is administered through repeated insufflation of an arterial pressure cuff in one of the patient arms, which in theory liberates vasoactive mediators that prevents the ischemic damage to the kidneys secondary to contrast media. All of the patients will receive endovenous normal saline to prevent nephropathy, which is a common strategy in our institution. Half of the patients will receive remote ischemic preconditioning while the other half will only receive a dummy preconditioning intended to keep the double blind strategy of the trial.

The main endpoint will be to ascertain the incidence of contrast induced nephropathy in both arms of the study, as a way to evaluate the efficacy of this strategy.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in general wards, emergency room or ambulatory consult.
* 18 years or older.
* Requires computerized tomography with endovenous contrast.
* Glomerular filtration rate between 30 - 60 mL/minute/1,73 m2.
* Patient accepts and signs informed consent.

Exclusion Criteria:

* Allergic to contrast media.
* Unable to accept or sign informed consent.
* Did not received endovenous saline before and/or after the contrast procedure.
* Peripheral arterial disease.
* Bilateral upper extremities lymph node dissection or any situation impending arterial pressure taking.
* Morbid obesity (body mass index 40 or more).
* Arterial systolic pressure greater than 175 mmHg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2018-10-09 (Actual)

PRIMARY OUTCOMES:
Contrast induced nephropathy incidence | 48 to 72 hours
  Increase in serum creatinine by 0,3 mg/dL compared to initial values.

SECONDARY OUTCOMES:
Adverse effects to preconditioning. | 0 to 72 hours.
  Any of pain in upper extremities, petechiae, bleeding from venopuncture sites, erythema.

CONTACTS AND LOCATIONS:
Locations (1):
- Grupo Nefrología Fundación Valle del Lili, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rudnick M, Feldman H. Contrast-induced nephropathy: what are the true clinical consequences? Clin J Am Soc Nephrol. 2008 Jan;3(1):263-72. doi: 10.2215/CJN.03690907. PMID 18178787
- [Background] Holscher B, Heitmeyer C, Fobker M, Breithardt G, Schaefer RM, Reinecke H. Predictors for contrast media-induced nephropathy and long-term survival: prospectively assessed data from the randomized controlled Dialysis-Versus-Diuresis (DVD) trial. Can J Cardiol. 2008 Nov;24(11):845-50. doi: 10.1016/s0828-282x(08)70193-4. PMID 18987758
- [Background] Goldenberg I, Matetzky S. Nephropathy induced by contrast media: pathogenesis, risk factors and preventive strategies. CMAJ. 2005 May 24;172(11):1461-71. doi: 10.1503/cmaj.1040847. PMID 15911862
- [Background] Bonventre JV. Limb ischemia protects against contrast-induced nephropathy. Circulation. 2012 Jul 24;126(4):384-7. doi: 10.1161/CIRCULATIONAHA.112.119701. Epub 2012 Jun 26. No abstract available. PMID 22735307
- [Background] Gassanov N, Nia AM, Caglayan E, Er F. Remote ischemic preconditioning and renoprotection: from myth to a novel therapeutic option? J Am Soc Nephrol. 2014 Feb;25(2):216-24. doi: 10.1681/ASN.2013070708. Epub 2013 Dec 5. PMID 24309187